CLINICAL TRIAL: NCT01888029
Title: Influence of Transcranial Direct Current Stimulation on Cortical Plasticity in Patients With Mild Cognitive Impairment (MCI)
Brief Title: Influence of tDCS on Cortical Plasticity in Patients With Mild Cognitive Impairment (MCI)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Plasticity in MCI
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Patients With Mild Cognitive Impairment
Keywords: mild cognitive impairment; Transcranial Direct Current Stimulation; Cortical Plasticity
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial direct current stimulation (Experimental)
  Interventions: Device: transcranial direct current stimulation
- sham stimulation (Placebo Comparator)
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation
  Arms: transcranial direct current stimulation
Device: sham stimulation
  Arms: sham stimulation

SUMMARY:
The aim of this study is to investigate whether the anodal transcranial direct current stimulation (tDCS) over the primary motor cortex (M1) in patients with mild cognitive impairment (MCI) leads to an increase in cortical plasticity (change in motor evoked potentials (MEP) in mV).

ELIGIBILITY:
Inclusion Criteria:

* Right-handed according to the Oldfield Händigkeits inventory (lateralization index> 70) (1971)
* Cognitive impairment according to the diagnostic criteria of a MCI (amnesic or even multiple domains)
* No therapeutic treatment with AChE inhibitors
* No motor impairments relevant to everyday life
* Age 50 to 80 years

Exclusion Criteria:

* Severe neurological / psychiatric or pre-existing internist conditions because additional cognitive deficits are expected
* Epilepsy, epileptic seizure in medical history
* Cognitive deficit (MMSE <20)
* Depressive episode (Beck Depression Inventory (BDI)> 12)
* Newly taking (<3 months) centrally active drugs, particularly acetylcholinesterase inhibitors
* Pregnancy
* Pacemaker (contraindication for MRI)
* Other metal parts in the body (contraindication for MRI)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the anodal transcranial direct current stimulation over the primary motor cortex (M1) in patients with mild cognitive impairment (MCI) | 1 week
  to investigate whether the anodal transcranial direct current stimulation over the primary motor cortex (M1) in patients with mild cognitive impairment (MCI) increases cortical plasticity (measured via motor evoked potentials) compared to sham stimulation

SECONDARY OUTCOMES:
Comparison of tDCS-induced changes on central cholinergic activity | 1 week
  to investigate weather the anodal transcranial direct current stimulation affect central cholinergic activity (measured via a TMS protocol) in MCI patients compared to sham stimulation
Comparison of tDCS-induced changes in learning success | 1 week
  tDCS-induced changes in learning success (performance in a motor learning paradigm in patients with MCI after tDCS vs. sham stimulation)
MR elastography | 1 week
  Comparison of viscoelastic parameters in cerebral MR elastography in patients with MCI
genetic polymorphism, ApoE4 | once
  optional assessment of genetic Apo4 epsilon status for assessment of differences in cortical plasticity and elasticity between Apo4 epsilon positive and negative participants

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Neurologie, Charité Universitätsmedizin Berlin, Berlin, Germany